CLINICAL TRIAL: NCT00406042
Title: The Role of Topical Prednisolone Acetate Following Selective Laser Trabeculoplasty
Brief Title: The Role of Steroids Following Selective Laser Trabeculoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16678
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2007-03-29 (Estimated); Status verified 2007-03

CONDITIONS: Glaucoma
Keywords: glaucoma; trabeculoplasty; steroids
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: prednisolone acetate 1%

SUMMARY:
To evaluate whether or not using topical steroids after selective laser trabeculoplasty affects intraocular pressure outcomes.

DETAILED DESCRIPTION:
Subjects undergoing bilateral SLT will be randomly assigned to use prednisolone acetate 1% in one eye four times daily with no treatment in the fellow eye, for one week following SLT. Examinations will occur at baseline, and one week, one month and three months after SLT. IOP and anterior chamber inflammation will be noted at each visit.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma or ocular hypertension
* need for bilateral SLT

Exclusion Criteria:

* eye disease precluding accurate IOP measurement
* contraindication to topical prednisolone acetate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2005-09; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure reduction

SECONDARY OUTCOMES:
Anterior chamber inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Tony Realini, MD, Principal Investigator — West Virginia University Eye Institute
Locations (1):
- West Virginia University Eye Institute, Morgantown, West Virginia, United States

REFERENCES:
- [Derived] Realini T, Charlton J, Hettlinger M. The impact of anti-inflammatory therapy on intraocular pressure reduction following selective laser trabeculoplasty. Ophthalmic Surg Lasers Imaging. 2010 Jan-Feb;41(1):100-3. doi: 10.3928/15428877-20091230-18. PMID 20128578